CLINICAL TRIAL: NCT03641872
Title: A Prospective Multi-center Validating Cohort for ACLF Diagnosis and Prognosis From Ch-CANONIC Study
Brief Title: A Validation Cohort for ACLF Diagnosis and Prognosis
Acronym: Ch-CANONIC-Val
Status: Completed | Type: Observational
Sponsor: Hai Li (Other)
Responsible Party: Sponsor-Investigator, Hai Li, Official Title: Professor, Department of Gastroenterology, RenJi Hospital ; Vice Director of the National Digestive Key Laboratory; Youth Commission of Chinese Society of Hepatology., Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: CHINA-ACLF-2
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Liver Failure, Acute on Chronic; Liver Dysfunction
Keywords: acute-on-chronic liver disease; acute decompensation; multiple organ failures; acute-on-chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Diseases; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute-on-Chronic Liver Disease: 1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients and non-alcoholic fatty liver disease patients.
  2. ALI(acute liver injury): including [ALT > 3 ULN(upper limited of normal),AST > 3 ULN or TB > 2 ULN within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy, bacterial infection, gastrointestinal bleeding and/or jaundice(TB > 5 ULN) within 1 month before enrollment)].
  3. Standary therapy for chronic liver disease with ATI and/or AD
  Interventions: Other: Standary therapy

INTERVENTIONS:
Other: Standary therapy — Standary therapy for chronic liver disease with ALI and/or AD

SUMMARY:
Acute on chronic liver failure (ACLF) is a distinct entity encompassing the acute deterioration of liver function, culminating in multiple organs failure and high short-term mortality. Definitions and descriptions of ACLF vary between Western and Eastern types, and alcoholism and hepatitis B virus (HBV) are the main etiologies, respectively. To determine whether there are unified diagnostic criteria, severity classification and prognostic model for different etiologies of ACLF. Investigators had launched a multicenter prospective cohort with the same inclusion criteria and disease indicators as those used in the European CANONIC (Chronic liver failure-ACLF in Cirrhosis) study in China，the Ch-CANONIC study(NCT02457637). From Jan 2015 to Dec 2016, 2,600 inpatients with chronic liver disease complicated with ALI and/or AD were recruited. Data were collected during a 28-day hospitalization and continuous follow-ups were performed once a month until 36 months after hospitalization (at least 18 months up to now). Of these patients, 71.5% had HBV-related disease, 1833 had cirrhotic disease, and 767 had non-cirrhotic disease diagnosed by CT scan.

Due to the lack of pathological gold standards, the diagnosis of ACLF is based on the clinical assessment of short-term mortality from organ functional parameters. In subsequent statistics and data analysis, investigators focused on (but not limit in) the relationship between short-term mortality and 6 parameters (bilirubin, INR, Creatinine, SpO2/FiO2, mean arterial pressure and West-Haven grade) from CLIF-C OFs (Chronic liver failure-Consortium Organ Failure score). And then a specific mathematical model has been constructed to obtain the available organ failure cutoff values. Subsequently, investigators carried out a diagnostical criteria for ACLF based on the results obtained from the model and get a good internal-validation result through risk ratio. Meanwhile, investigators conducted a precise prediction model for patients' prognosis and achieved a good predictive effect with consistency by AUC internal-validation. In addition, investigators summarized the course and some characteristics of ACLF.

Therefore, investigators hope to launch another prospective multi-center cohort study with the same inclusion and exclusion criteria, and continue to recruit 800 to 900 patients (about 30% of the previous cohort) as the external validation cohort for the preliminary results mentioned above.

DETAILED DESCRIPTION:
Acute-on chronic liver failure (ACLF) was first described by Japanese researchers in 1995. In 2011, the American Association for the Study of Liver Disease (AASLD) and the European Association for the Study of the Liver (EASL) concluded that the core characteristics of ACLF were multiple organ failures and high short-term mortality. In 2013, the EASL-CLIF (the European Association for the Study of The Liver-chronic liver failure) established the CLIF-SOFA (chronic liver failure-sequential organ failure assessment) criteria of ACLF through a prospective multicenter study at 29 liver units in eight European countries for 1 year, with a focus on patients with alcoholic cirrhosis with acute decompensation (AD). In the Asia-Pacific region, the majority of liver disease is viral hepatitis, while in western countries, it is alcoholic liver disease. There is a sharp east-west divide with respect to the definition of ACLF, especially in the definition of chronic liver disease and related organ failure.

In 2014, investigators had analyzed 6 years' data of hepatitis B virus (HBV)-related chronic liver disease in patients with AD in two affiliated hospitals of Shanghai Jiao Tong University School of Medicine. These data were also quantified and sent to the EASL-CLIF center for analysis. 80% of whole patients were clinically diagnosed with cirrhosis, 30% of which had pathological diagnosis. Through analysis of the liver tissues of the liver transplantation (LT) patients, 95% had pseudo-lobules. The residual 5% of liver tissues were in the S3 stage of progressive liver fibrosis. Moreover, the research also demonstrated that the pathological characteristics of ACLF may be MHN/SMHN (massive hepatic necrosis/submassive hepatic necrosis) in the background of liver pseudo-lobules. Regeneration of hepatic progenitor cells, cholestasis, and sepsis are other possible pathological features of ACLF.

Compared with the CANONIC (EASL-CLIF Acute-on-Chronic Liver Failure in Cirrhosis), there are many similarities between ACLF patients with alcoholic cirrhosis or HBV induced cirrhosis.But ACLF patients with cirrhosis induced by HBV or alcoholism differ in main types of organ failure. According to CLIF-C OFs (CLIF-C organ failure score), the incidence of 6 organ failures is not exactly the same in the two types of ACLF. Even for the same type of organ failure, the short-term mortality of patients is different.

To determine whether there are unified diagnostic criteria, disease grades classification and prognostic model for different etiologies of ACLF, Investigators had launched a multicenter prospective cohort with the same inclusion criteria and disease indicators as those used in the European CANONIC study in China，the Ch-CANONIC study (NCT02457637). The research was carried out in 14 Chinese national wide liver centers each of whose total beds are around 500. From Jan 2015 to Dec 2016, 2600 inpatients with chronic liver disease (including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis, non-alcoholic fatty liver disease or alcoholic liver disease patients) complicated with AD [acute decompensation): including [(having ascites, hepatic encephalopathy, bacterial infection, gastrointestinal bleeding or jaundice (TB>5NL) within 1 month before enrollment] and/or ALI [acute liver injury: including ALT>3NL (normal level), AST>3NL or TB>2NL within 1 week before enrollment] were recruited. Data were collected during a 28-day hospitalization and continuous follow-ups were performed once a month until 36 months after hospital discharge. Of these patients, 71.5% (1859/2600) had HBV-related disease,71.5% (1833/2600) had cirrhotic disease, and 28.5% (767/2600) had non-cirrhotic disease.

Up to now, every recruited patient has been followed-up for at least 18 months. Thus, a large amount of data has been collected for analysis. The preliminary results of our research are as follows (As the relevant papers are being reviewed, the detailed data will be updated in subsequent protocols):

1. Investigators explored the epidemiology of inpatients with severe chronic liver disease and the risk of high short-term mortality in nationwide hospitals, including the prevalence of acute deterioration, the disease burden and the clinical features of patients with short-term mortality.
2. Investigators had got some conclusions from many observations of the clinical course of patients with short-term mortality. The time interval from acute insults to different endpoints, including AD, organ failure and death was carefully evaluated. Moreover, the distribution and regularity of mortality within a one-year follow-up had also been plotted.
3. Due to the lack of pathological gold standards, the diagnosis of ACLF is based on the clinical assessment of short-term mortality from organ functional parameters. Investigators implemented a statistical approach to determine cut-off values for vital organ damage and failure. In subsequent statistics and data analysis, refer to the CANONIC study, at the beginning investigators focused on (but not limit in) the relationship between short-term mortality and 6 parameters (bilirubin, International Normalized Ratio, Creatinine, SpO2/FiO2, mean arterial pressure and West-Haven grade) from CLIF-C OFs. And then a specific an evidence-based model has been constructed to obtain the available organ failure cutoff values. Subsequently, investigators established a diagnostical criteria for ACLF based on the results obtained from the model to quantify the severity of the disease.
4. A prognosis model was established to define high disease risk patients to distinguish early-stage ACLF patients (pre-ACLF) from non-ACLF patients with AD or ALI. Investigators achieved a good predictive effect with consistency by AUC internal-validation.
5. Implementation of high-throughput screening by proteomic and metabolomic studies to screen and validate biomarkers for the prediction of ACLF in the early stage and establish a prognostic evaluation for ACLF using plasma from a biobank; execution of a Genome-wide Association Study (GWAS) using DNA samples extracted from peripheral blood mononuclear cells; and exploration of the mechanism of ACLF disease progression by studying DNA levels (GWAS), protein levels (proteomic analysis) and metabolite levels (metabolomic analysis). This part of work is in progress.

Therefore, investigators hope to launch another cohort study with the same inclusion/exclusion criteria and recruit 800-900 patients (about 30% of the previous cohort) as the external validation cohort for the preliminary results (1~4) mentioned above.

Overall, 800-900 inpatients will be enrolled continuously from Sep. 2018 to Mar. 2019(anticipated). The research will be carried out in about 12 Chinese national wide liver centers each of whose total beds are around 500. Every patient will have a unique number. Cirrhosis or non-cirrhosis will be diagnosed by CT, FibroScan and FIB-4 index. The investigators will take the note of the history of their liver disease and find the etiology of their liver disease, such as hepatitis B, NAFLD, alcoholic liver disease, and autoimmune liver disease. For viral hepatitis, the investigators will ask how antiviral therapy is conducted. The investigators will ascertain if the patients have a history of cirrhosis and for how long. The investigators will ascertain if the patients have any of the following predisposing factors: HBV reactivation, bacterial infection, active alcohol intake, HBV superimposed by other hepatitis viruses, gastrointestinal bleeding, portal vein thrombosis, surgery, intake of hepatotoxic drugs or herbs, or physiological exhaustion. The investigators will establish the main cause of admission: gastrointestinal bleeding, hepatic encephalopathy, ascites, bacterial infection, jaundice or ALI. The investigators will determine whether the patients have chronic disease such as hypertension, coronary heart disease, diabetes, chronic renal disease, or connective tissue disease.

During hospitalization, data will be collected at 1, 7,14, 21 and 28 days (or last visit date, if the patient is hospitalized less than 28 days), and 24h prior to death or LT (if the patient dies or has LT) and focus on the following three aspects.

The first aspect is evaluation of organ failure. The circulatory system will be evaluated by measuring heart rate and blood pressure and use of vasopressors. Renal function will be evaluated by serum creatinine or renal replacement therapy. Coagulation function will be evaluated by INR (international normalized ratio of prothrombin time). Liver function will be evaluated by serum total bilirubin. The respiratory system will be evaluated by the oxygenation index (SpO2/FiO2), and whether the patient needs nasal catheter oxygen and artificial ventilation will also be recorded. The nervous system will be evaluated by the West-Haven grade of hepatic encephalopathy. Bacterial infection, including pneumonia, urinary tract infection, spontaneous bacterial peritonitis, spontaneous bacteremia, and cellulitis will be evaluated by positive culture results or imaging findings.The investigators will establish whether ascites and hepatic encephalopathy can be medically controlled.

The second aspect is laboratory examinations. Tests at admission will include routine blood, urine and stool tests, liver and renal function tests, blood electrolytes, blood-gas analysis, blood glucose, coagulation test, C-reactive protein (CRP), procalcitonin (PCT), HBV antibodies and antigens, anti-hepatitis A (IgM), HBV-DNA, anti-hepatitis E (IgM), anti-hepatitis C, and immunoglobulins (IgA, IgG, IgM and IgM-4). Tests at other times will include blood, urine and stool routine tests, liver and renal function tests, blood electrolytes, blood glucose, coagulation test, CRP (C-reactive protein) and PCT (procalcitonin). Tests optionally done during hospitalization will include autoantibody measurement. Blood，sputum，ascites culture or middle urine cultivation will be taken if a patient is suspected of having a relevant infection.

The third aspect is imaging. During hospitalization, thoracic X ray or computed tomography (CT) will be done to diagnose pulmonary infection. Abdominal CT (enhanced when necessary), B ultrasound and FibroScan or other elastography will be done to diagnose cirrhosis (or fibrosis), portal thrombosis, esophageal and gastric varices and hepatocellular carcinoma.

Follow-up will be clinical visiting, but telephone call will be acceptable for patients unable to attend. Clinical follow-up is once a month for 3 months adding to 3 visits. Laboratory tests should be taken at least once (the last visit is perferred) including routine blood tests, liver and renal function test, coagulation test, CRP and PCT. B ultrasound will be done to monitor cirrhosis (or fibrosis) , complications and hepatocellular carcinoma. During follow-up, patients will be hospitalized again whenever they have new ALI or AD. Similar data will be collected reference to their prior admission and follow-up will restart. If the patients die during follow-up, the time of death and main cause of death will be noted. When the patients undergo LT during follow-up, the time of LT and the results of hepatic pathology will be noted.

Demographic data, disease history, baseline data after admission and follow-up data after discharge will be recorded in a similar process and quality control. But investigators plan to simplify some data collection work. Concretely, (1) During hospitalization, data will be recorded and followed up once a week (but must include the first and last day's data of hospitalization).(2) Samples of feces and urine are no longer collected. (3) The duration of follow-up for each discharged patient will be shorten from 36 months to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* inpatient (hospitalization >1 days)(including patient in emergency observation wards)chronic liver disease patients including non-alcoholic fatty liver disease patients,chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients and decompensated cirrhosis patients
* having acute liver injury [ALT(alanine aminotransferase)>3ULN,AST(aspartate aminotransferase)>3ULN or TB(total bilirubin)>2 ULN within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy, bacterial infection ,gastrointestinal bleeding or jaundice(TB>5NL)within 1 month before enrollment].

Exclusion Criteria:

* pregnancy
* hepatocellular carcinoma or other liver malignancies
* malignancy of other organs
* severe chronic extrahepatic disease including chronic obstructive pulmonary disease combined with respiratory failure, coronary heart disease with cardiac function level 3 (NYHA), myocardial infarction in the 3 months before admission, diabetes with severe complications and chronic kidney disease with end-stage renal failure receiving immunosuppressive drugs for reasons other than chronic liver disease

Ages: 15 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chronic liver disease patients（with liver dysfunction more than 6 months） with acute liver injury[with ALT>3 ULN),AST>3NL or TB>2 ULN within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy, bacterial infection ,gastrointestinal bleeding or jaundice(TB > 5ULN)within 1 month before enrollment].
Sampling Method: Probability Sample
Enrollment: 1370 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Short-Term Mortality & | Up to 3 months
  Mortality will be calculated and reported at 28 days,90 days.
Short-Term Liver Transplantation Rate | Up to 3 months
  Liver Transplantation Rate will be calculated and reported at 28 days,90 days.Those who undergoing liver transplantation are patients developed life-threatening liver failure. If those patients do not got a chance of transplantation, there would be a high probability that they could die in a very short period of time.So Liver Transplantation Rate is also a Primary Outcome Measure.

SECONDARY OUTCOMES:
the Appearance of liver failure | Up to 28 days
  The appearance of liver failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
the Appearance of coagulation failure | Up to 28 days
  The appearance of coagulation failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
the Appearance of renal failure | Up to 28 days
  The appearance of renal failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
the Appearance of circulative failure | Up to 28 days
  The appearance of circulative failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
the Appearance of CNS failure | Up to 28 days
  The appearance of respiratory failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
the Appearance of respiratory failure | Up to 28 days
  The appearance of respiratory failure will be evaluated and reported at the 1st day, once a week and last visit during patients' hospitalization.
Serum bilirubin | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
International Normalized Ratio(INR) | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
Serum creatinine | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
Aminotransferase | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
Alkaline phosphatase(AKP) | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
γ-Glutamyltransferase(γ-GT) | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.
white blood cell count/neutrophil count | Up to 28 days
  The biochemical parameter will be collected and reported at the 1st day, once a week and last visit during patients' hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, Study Director — Digestive Department of Renji Hospital,Shanghai Jiao Tong University School of Medicine
Locations (12):
- China (12):
  - Ditan Hospital of integrated traditional Chinese and Western Medicine Center, Beijing, Beijing Municipality
  - Southwest Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Southern hospital infection department, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Wuhan Union Hospital of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Renji hospital of Shanghai Jiao Tong University School of Medical, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Infectious Disease Center, The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gu WY, Xu BY, Zheng X, Chen J, Wang XB, Huang Y, Gao YH, Meng ZJ, Qian ZP, Liu F, Lu XB, Shang J, Li H, Wang SY, Sun X, Li H. Acute-on-Chronic Liver Failure in China: Rationale for Developing a Patient Registry and Baseline Characteristics. Am J Epidemiol. 2018 Sep 1;187(9):1829-1839. doi: 10.1093/aje/kwy083. PMID 29762630
- [Background] Ohnishi H, Sugihara J, Moriwaki H, Muto Y. [Acute-on-chronic liver failure]. Ryoikibetsu Shokogun Shirizu. 1995;(7):217-9. No abstract available. Japanese. PMID 8749457
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Kamath PS, Kim WR; Advanced Liver Disease Study Group. The model for end-stage liver disease (MELD). Hepatology. 2007 Mar;45(3):797-805. doi: 10.1002/hep.21563. PMID 17326206
- [Background] Vallet-Pichard A, Mallet V, Nalpas B, Verkarre V, Nalpas A, Dhalluin-Venier V, Fontaine H, Pol S. FIB-4: an inexpensive and accurate marker of fibrosis in HCV infection. comparison with liver biopsy and fibrotest. Hepatology. 2007 Jul;46(1):32-6. doi: 10.1002/hep.21669. PMID 17567829
- [Background] Sarin SK, Kumar A, Almeida JA, Chawla YK, Fan ST, Garg H, de Silva HJ, Hamid SS, Jalan R, Komolmit P, Lau GK, Liu Q, Madan K, Mohamed R, Ning Q, Rahman S, Rastogi A, Riordan SM, Sakhuja P, Samuel D, Shah S, Sharma BC, Sharma P, Takikawa Y, Thapa BR, Wai CT, Yuen MF. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific Association for the study of the liver (APASL). Hepatol Int. 2009 Mar;3(1):269-82. doi: 10.1007/s12072-008-9106-x. Epub 2008 Nov 20. PMID 19669378
- [Background] Bajaj JS, O'Leary JG, Reddy KR, Wong F, Biggins SW, Patton H, Fallon MB, Garcia-Tsao G, Maliakkal B, Malik R, Subramanian RM, Thacker LR, Kamath PS; North American Consortium For The Study Of End-Stage Liver Disease (NACSELD). Survival in infection-related acute-on-chronic liver failure is defined by extrahepatic organ failures. Hepatology. 2014 Jul;60(1):250-6. doi: 10.1002/hep.27077. Epub 2014 May 29. PMID 24677131
- [Background] Jalan R, Saliba F, Pavesi M, Amoros A, Moreau R, Gines P, Levesque E, Durand F, Angeli P, Caraceni P, Hopf C, Alessandria C, Rodriguez E, Solis-Munoz P, Laleman W, Trebicka J, Zeuzem S, Gustot T, Mookerjee R, Elkrief L, Soriano G, Cordoba J, Morando F, Gerbes A, Agarwal B, Samuel D, Bernardi M, Arroyo V; CANONIC study investigators of the EASL-CLIF Consortium. Development and validation of a prognostic score to predict mortality in patients with acute-on-chronic liver failure. J Hepatol. 2014 Nov;61(5):1038-47. doi: 10.1016/j.jhep.2014.06.012. Epub 2014 Jun 17. PMID 24950482
- [Background] Sarin SK, Kedarisetty CK, Abbas Z, Amarapurkar D, Bihari C, Chan AC, Chawla YK, Dokmeci AK, Garg H, Ghazinyan H, Hamid S, Kim DJ, Komolmit P, Lata S, Lee GH, Lesmana LA, Mahtab M, Maiwall R, Moreau R, Ning Q, Pamecha V, Payawal DA, Rastogi A, Rahman S, Rela M, Saraya A, Samuel D, Saraswat V, Shah S, Shiha G, Sharma BC, Sharma MK, Sharma K, Butt AS, Tan SS, Vashishtha C, Wani ZA, Yuen MF, Yokosuka O; APASL ACLF Working Party. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific Association for the Study of the Liver (APASL) 2014. Hepatol Int. 2014 Oct;8(4):453-71. doi: 10.1007/s12072-014-9580-2. Epub 2014 Sep 26. PMID 26202751
- [Background] Arroyo V, Moreau R, Jalan R, Gines P; EASL-CLIF Consortium CANONIC Study. Acute-on-chronic liver failure: A new syndrome that will re-classify cirrhosis. J Hepatol. 2015 Apr;62(1 Suppl):S131-43. doi: 10.1016/j.jhep.2014.11.045. PMID 25920082
- [Background] Li H, Xia Q, Zeng B, Li ST, Liu H, Li Q, Li J, Yang SY, Dong XJ, Gao T, Munker S, Liu Y, Liebe R, Xue F, Li QG, Chen XS, Liu Q, Zeng H, Wang JY, Xie Q, Meng QH, Wang JF, Mertens PR, Lammert F, Singer MV, Dooley S, Ebert MP, Qiu DK, Wang TL, Weng HL. Submassive hepatic necrosis distinguishes HBV-associated acute on chronic liver failure from cirrhotic patients with acute decompensation. J Hepatol. 2015 Jul;63(1):50-9. doi: 10.1016/j.jhep.2015.01.029. Epub 2015 Jan 31. PMID 25646889
- [Background] Li H, Chen LY, Zhang NN, Li ST, Zeng B, Pavesi M, Amoros A, Mookerjee RP, Xia Q, Xue F, Ma X, Hua J, Sheng L, Qiu DK, Xie Q, Foster GR, Dusheiko G, Moreau R, Gines P, Arroyo V, Jalan R. Characteristics, Diagnosis and Prognosis of Acute-on-Chronic Liver Failure in Cirrhosis Associated to Hepatitis B. Sci Rep. 2016 May 5;6:25487. doi: 10.1038/srep25487. PMID 27146801
- [Background] Hernaez R, Sola E, Moreau R, Gines P. Acute-on-chronic liver failure: an update. Gut. 2017 Mar;66(3):541-553. doi: 10.1136/gutjnl-2016-312670. Epub 2017 Jan 4. PMID 28053053
- [Background] Dusheiko G, Agarwal K. Delineating the global challenges of hepatitis B virus infection. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):372-373. doi: 10.1016/S2468-1253(18)30093-1. Epub 2018 Mar 27. No abstract available. PMID 29599077
- [Background] Deboeck PR, Nicholson J, Kouros C, Little TD, Garber J. Integrating developmental theory and methodology: Using derivatives to articulate change theories, models, and inferences. Appl Dev Sci. 2016;19(4):217-231. doi: 10.1080/10888691.2015.1021924. PMID 26949327
- [Derived] Zhang Y, Tan W, Wang X, Zheng X, Huang Y, Li B, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Shi Y, Shang J, Yan H, Zheng Y, Zhang W, Gu W, Qiao L, Deng G, Zhou Y, Hou Y, Zhang Q, Xiong S, Liu J, Duan L, Chen R, Chen J, Jiang X, Luo S, Chen Y, Jiang C, Zhao J, Ji L, Mei X, Li J, Li T, Zheng R, Zhou X, Ren H, Cheng X, Guo L, Li H; Chinese (Acute on) Chronic Liver Failure Consortium (Ch-CLIF.C). Metabolic biomarkers significantly enhance the prediction of HBV-related ACLF occurrence and outcomes. J Hepatol. 2023 Nov;79(5):1159-1171. doi: 10.1016/j.jhep.2023.07.011. Epub 2023 Jul 29. PMID 37517452
- [Derived] Wang T, Tan W, Wang X, Zheng X, Huang Y, Li B, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Yan H, Zheng Y, Zhang W, Yin S, Gu W, Zhang Y, Dong F, Wei J, Deng G, Xiang X, Zhou Y, Hou Y, Zhang Q, Xiong S, Liu J, Long L, Chen R, Chen J, Jiang X, Luo S, Chen Y, Jiang C, Zhao J, Ji L, Mei X, Li J, Li T, Zheng R, Zhou X, Ren H, Shi Y, Li H; Chinese (Acute on) Chronic Liver Failure Consortium (Ch-CLIF.C). Role of precipitants in transition of acute decompensation to acute-on-chronic liver failure in patients with HBV-related cirrhosis. JHEP Rep. 2022 Jul 5;4(10):100529. doi: 10.1016/j.jhepr.2022.100529. eCollection 2022 Oct. PMID 36052222
- [Derived] Mei X, Li H, Deng G, Wang X, Zheng X, Huang Y, Chen J, Meng Z, Gao Y, Liu F, Lu X, Shi Y, Zheng Y, Yan H, Zhang W, Qiao L, Gu W, Zhang Y, Xiang X, Zhou Y, Sun S, Hou Y, Zhang Q, Xiong Y, Zou C, Chen J, Huang Z, Li B, Jiang X, Zhong G, Wang H, Chen Y, Luo S, Gao N, Liu C, Li J, Li T, Zheng R, Zhou X, Ren H, Yuan W, Qian Z. Prevalence and clinical significance of serum sodium variability in patients with acute-on-chronic liver diseases: a prospective multicenter study in China. Hepatol Int. 2022 Feb;16(1):183-194. doi: 10.1007/s12072-021-10282-8. Epub 2022 Jan 17. PMID 35037228
- [Derived] Ouyang R, Li H, Xia J, Wang X, Zheng X, Huang Y, Meng Z, Gao Y, Qian Z, Liu F, Lu X, Shi Y, Shang J, Liu J, Deng G, Zheng Y, Yan H, Zhang W, Qiao L, Jiang X, Wang H, Zhong G, Li B, Chen J. Lower platelet counts were associated with 90-day adverse outcomes in acute-on-chronic liver disease patients. Ann Palliat Med. 2021 Sep;10(9):9342-9353. doi: 10.21037/apm-21-1019. Epub 2021 Aug 13. PMID 34412498
- [Derived] Qiao L, Wang X, Deng G, Huang Y, Chen J, Meng Z, Zheng X, Shi Y, Qian Z, Liu F, Gao Y, Lu X, Liu J, Gu W, Zhang Y, Wang T, Wu D, Dong F, Sun X, Li H. Cohort profile: a multicentre prospective validation cohort of the Chinese Acute-on-Chronic Liver Failure (CATCH-LIFE) study. BMJ Open. 2021 Jan 8;11(1):e037793. doi: 10.1136/bmjopen-2020-037793. PMID 33419900
- [Derived] Zhang Y, Xu BY, Wang XB, Zheng X, Huang Y, Chen J, Meng ZJ, Gao YH, Qian ZP, Liu F, Lu XB, Shi Y, Shang J, Li H, Wang SY, Yin S, Sun SN, Hou YX, Xiong Y, Chen J, Li BL, Lei Q, Gao N, Ji LJ, Li J, Jie FR, Zhao RH, Liu JP, Lin TF, Chen LY, Tan WT, Zhang Q, Zou CC, Huang ZB, Jiang XH, Luo S, Liu CY, Zhang YY, Li T, Ren HT, Wang SJ, Deng GH, Xiong SE, Liu XX, Wang C, Yuan W, Gu WY, Qiao L, Wang TY, Wu DD, Dong FC, Li H, Hua J. Prevalence and Clinical Significance of Portal Vein Thrombosis in Patients With Cirrhosis and Acute Decompensation. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2564-2572.e1. doi: 10.1016/j.cgh.2020.02.037. Epub 2020 Feb 25. PMID 32109631